CLINICAL TRIAL: NCT03652103
Title: Efficiency of Erector Spinae Plane Block For Patients Undergoing Percutaneous Nephrolithotomy: A Prospective, Randomized, Controlled, Single Blind Study
Brief Title: Efficiency of Erector Spinae Plane Block For Patients Undergoing Percutaneous Nephrolithotomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mehmet Uğur Bilgin, Anesthesiology Resident, Bozyaka Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESPforPNL
Record Dates: First submitted 2018-08-28; First posted 2018-08-29 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Nephrolithotomy, Percutaneous; Anesthetics, Local; Nerve Block; Erector Spinae Plane Block; Pain, Postoperative; Anesthesia and Analgesia
Keywords: Truncal Nerve Blocks, Ultrasound Guided Nerve Blocks
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Two groups involved. First group will receive total intravenous anesthesia and erector spinae plane block catheter Second group will receive total intravenous anesthesia and routine analgesia protocol for percutaneous Nephrolithotomy procedures.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GCont (No Intervention): Only dressing will be applied to patients without actually nerve catheter performed
- GBlock (Experimental): Ultrasound Guided Erector Spinae Plane Block Catheter will be applied: 20ml Bupivacaine 0.25% Injectable Solution* will be administered initially.
  20 ml Bupivacaine %0.25 Injectable Solution** will be administered 30 minutes before ambulation at postoperative day(POD) 0 and before removal of nephrostomy at POD 2
  *10ml %0,5 Bupivacaine will be diluted with 10ml Saline solution.
  Interventions: Procedure: Ultrasound Guided Erector Spinae Plane Block Catheterisation; Drug: Bupivacaine 0.25% Injectable Solution

INTERVENTIONS:
Procedure: Ultrasound Guided Erector Spinae Plane Block Catheterisation — After receiving general anesthesia, patients will positioned prone. Before operation begins, ESP block catheter will be applied with ultrasound guidance to the same level as surgeon's incision.
  Arms: GBlock
Drug: Bupivacaine 0.25% Injectable Solution — Perineural Injection
  Other Names: Marcain
  Arms: GBlock

SUMMARY:
Investigators' goal is to determine whether Erector Spinae Plane Block would provide a better analgesia, help mobilization and early discharge or increase satisfaction for patients undergoing Percutaneous Nephrolithotomy(PNL).

One of the two groups will receive ESP catheterization after general anesthesia conducted. The other group will receive routine analgesia protocol used for PNL.

The total amount of drugs administered, pain scores(NRS) at certain time intervals and at certain events(removal of nephrostomy and pain at mobilization) will be recorded and compared.

DETAILED DESCRIPTION:
Erector Spinae Plane Block(ESP) is a rather new method which can block ventral and dorsal rami of spinal nerves in the paravertebral area after they leave the spinal column. Originally used for thoracic somites, by spreading in a craniocaudal fashion in the erector spinae muscle group, it has the potential of blocking cervical or lumbar nerves as well.

To provide better analgesia for surgical procedures, anesthesiologists use truncal blocks for peripheral intervention. Although these blocks are generally very effective and easy to apply, they are limited by a relatively small area of effectivity. In order to achieve denser effects for larger surfaces, epidural anesthesia must be used with the risk of more severe complications than any peripheral or truncal nerve blocks. Epidural anesthesia also has the disadvantages of requiring more experience and more cautiousness than ultrasound-guided truncal blocks and risks of an undesirable temporary motor blockade. ESP block could be the answer for better regional analgesia while avoiding motor blockade and complications of epidural anesthesia.

The study will have two groups as Block Group(GB) and Control Group(GC) and two periods as during operation and 48 hours after the operation. Every participant will receive Total Intravenous Anesthesia(TIVA) and will be monitored with ECG, non-invasive blood pressure, heart rate, pulse oximeter, and Bispectral Index. Participants in GB will receive ultrasound-guided ESP block catheter after proper maintenance of anesthesia provided. The first period will be during operation. We will evaluate the administered drug amounts per kilogram for each patient. Investigators believe ESP block will help them deliver proper anesthesia with lower dosages. The second period will include postoperative 48 hours. Pain scores(NRS) will be evaluated at certain time intervals and at two critical moments between the two groups. One of the critical moment which patients fear and feel the pain most is the removal time of nephrostomy. The second moment is the first time patients start walking.

Rescue analgesia will be ordered on demand for both groups as IV 1 mg/kg tramadol. Hours and amounts of rescue analgesia administered will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for percutaneous nephrolithotomy under total intravenous anesthesia
* Patients who has informed consent for study
* Patients with American Society of Anesthesiologists Physical Status Classification(ASA) I and II

Exclusion Criteria:

* Patient's refusal to participate
* Patients under 18 years of age
* Patients who are undergoing surgery with an anesthesia technique other than total intravenous anesthesia for any reason (inhalation anesthesia, laryngeal mask application, etc.)
* Patients with known local anesthetic allergy
* Patients with Body mass index > 35
* Patients diagnosed sepsis and bacteriemia,
* Skin infection at the injection site,
* Patients with previous spinal surgery
* History of coagulopathy or anticoagulant therapy
* Patients with uncontrolled diabetes ,
* Uncoordinated patients,
* Psychological and emotional lability,
* Surgical intervention longer than 3 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2019-03-10 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Dosage of Drugs | During procedure
  Amounts of drugs per kilogram per hour will be recorded
Post-operative pain assessed by Numeric Rating Scale (NRS) | 30th minute postoperatively
  Pain scores will be recorded as reported by the patient according to NRS
Post-operative pain assessed by Numeric Rating Scale (NRS) | 60th minute postoperatively
  Pain scores will be recorded as reported by the patient according to NRS
Post-operative pain assessed by Numeric Rating Scale (NRS) | 2nd hour postoperatively
  Pain scores will be recorded as reported by the patient according to NRS
Post-operative pain assessed by Numeric Rating Scale (NRS) | 6th hour postoperatively
  Pain scores will be recorded as reported by the patient according to NRS
Post-operative pain assessed by Numeric Rating Scale (NRS) | 12th hour postoperatively
  Pain scores will be recorded as reported by the patient according to NRS
Post-operative pain assessed by Numeric Rating Scale (NRS) | 24th hour postoperatively
  Pain scores will be recorded as reported by the patient according to NRS
Post-operative pain assessed by Numeric Rating Scale (NRS) | 48th hour postoperatively
  Pain scores will be recorded as reported by the patient according to NRS
Post-operative pain assessed by Numeric Rating Scale (NRS) | Mobilisation at postoperative day (POD) 1
  Pain scores will be recorded during the first steps as reported by the patient according to NRS
Post-operative pain assessed by Numeric Rating Scale (NRS) | At the time of removal of nephrostomy at postoperative day (POD) 2
  Pain scores will be recorded during the procedure as reported by the patient according to NRS

SECONDARY OUTCOMES:
Opioid Consumption | 48 hour post-operatively
  Opioids(Tramadol) will be administered to patients in case demanded.
Discharge | 240 hours post-operatively
  Day of the discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Bozyaka Training and Research Hospital, Karabağlar, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No